CLINICAL TRIAL: NCT05885685
Title: Investigating the Effects of Nabilone on Endocannabinoid Metabolism in the Human Brain
Brief Title: Investigating the Effects of Nabilone on Endocannabinoid Metabolism
Acronym: NABI
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 098-2017; CAMHPET-CTA-109 (Other: CAMH)
Record Dates: First submitted 2023-05-23; First posted 2023-06-02 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Healthy
Keywords: nabilone; positron emission tomography
MeSH Terms: interventions — nabilone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Healthy Participants (Experimental): Participants will be prescribed a 1 week daily oral dose of nabilone which will begin at 0.25 mg and work their way up to 2 mg over the course of 7 days.
  Interventions: Drug: Nabilone Oral Capsule

INTERVENTIONS:
Drug: Nabilone Oral Capsule — Each oral capsule contains a 0.25 mg dose of nabilone. Participants begin by taking 1 capsule at night then 1 capsule in the morning and 1 at night for the next 2 days. On the 4th day, the dose is doubled. On the 6th day, the dose is doubled again.
  Other Names: TEVA-nabilone

SUMMARY:
The purpose of this study is to learn about the effects of a cannabis-like substance, nabilone, on the levels of endocannabinoid enzyme fatty acid amide hydrolase (FAAH) in brain of healthy individuals. Using magnetic resonance imagine (MRI) and positron emission tomography (PET), the main questions we aim to answer are: 1) Does nabilone decrease levels of FAAH in the brain? and 2) Are changes in levels of FAAH associated with clinical response to nabilone? Participants will complete:

* An in-person interview (~4 hours)
* Two brain imaging scanning sessions (~11 hours)
* A one week 2 mg titrated dose of nabilone
* Virtual check-ins (up to ~1.5 hours)

DETAILED DESCRIPTION:
There is limited data regarding the effect of exogenous cannabinoids, such as tetrahydrocannabinol (THC), on the endogenous cannabinoid system (eCS). Specifically, we do not know whether brain levels of fatty acid amide hydrolase (FAAH), the catabolic enzyme for the endocannabinoid anandamide, is affected by sub-chronic THC exposure.

Our primary objective is to use positron emission tomography (PET) imaging of the FAAH probe [11C]CURB to test the hypothesis that exposure to nabilone, a synthetic THC analogue, will reduce FAAH levels in the brain. Our secondary objective is to investigate whether reductions in FAAH levels are related to clinical response to nabilone.

Participant eligibility will be assessed through a series of questionnaires and assessments on medical, family, psychiatric and alcohol and drug use history. Individuals will also be required to provide blood and urine samples which we will test for recent drug use and pregnancy in female participants. Thirty healthy participants will complete one magnetic resonance imaging scan and two PET scans with [11C]CURB: one at baseline prior to nabilone administration and one approximately 4 weeks apart following a one week, 2 mg titrated dose of nabilone. Venous and arterial blood draws will be done during PET scans to measure FAAH genotype and plasma radiometabolites, respectively. Mood assessments will also be administered at these visits. During the nabilone dosing period, we will meet virtually with participants to check-in and monitor their tolerance and compliance.

Understanding whether recent nabilone exposure affects FAAH levels in brain may help to explain variability in clinical response to THC, the main psychoactive component in cannabis. This information can help guide therapeutic use of cannabis and cannabinoid derivatives, and aid in the development of evidence-based medicine targeting the eCS.

ELIGIBILITY:
Inclusion Criteria:

* Aged 19-65 years old. For safety reasons, we will ask participants to provide photo ID showing birthdate, in order to verify age.
* The ability to tolerate complete dosing regimen of nabilone (2mg titrated, 1 week course)
* Able to sign and date informed consent form.
* Willing and able to complete study as described in protocol

Exclusion Criteria:

* Serious, unstable medical condition including but not limited to cerebrovascular, renal, hepatic and coronary heart disease;
* Coagulation/Blood Disorders or use of anticoagulant medication
* Past or current neurological illness or head trauma;
* Lifetime diagnosis of DSM-5 Axis I psychiatric conditions including mood, anxiety, eating, somatoform and/or psychotic disorders and substance abuse and/or dependence;
* Suicidality or history of suicide attempts;
* Family history of psychotic disorders (first degree relative with a psychotic disorder);
* Current use (~30 days) of drugs of abuse that may affect the CNS, including cannabis;
* Tobacco dependence (Fagerstrom Test for Nicotine Dependence >4);
* Pregnancy or breastfeeding;
* Presence of metal objects in the body or implanted electronic devices, that preclude safe MR scanning;
* Claustrophobia;
* Known sensitivity to marijuana or other cannabinoid agents;
* Are on medications known to interact with nabilone such as: diazepam, sodium secobarbital, alcohol, codeine, any medications that affect mental and/or psychomotor function;
* Positive during drug screening for drugs of abuse;
* Exposure to radiation <20 mSv in the last 12 months and a number of PET scans that, including the number of PET scans under this protocol, will bring the total to more than 8 PET scans/lifetime, exceeding permissible limit for subjects participating in research set by Brain Health Imaging Centre Guideline;
* Participant has any other problem that, in the investigators opinion, would preclude participation in the trial;

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-10-31 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
[11C]CURB binding in the brain | 4 weeks
  Change in levels of [11C]CURB binding in the brain as indicated by the lambda k3 value from baseline to post-nabilone

SECONDARY OUTCOMES:
[11C]CURB decreases related to mood related assessments | 4 weeks
  Changes in mood related assessment Profile of Mood States (POMS) scores from baseline to post-nabilone. Negative subscales include tension (9 items, range 0-36), depression (15 items, range 0-60), fatigue (7 items, 0-28), confusion (7 items, range 0-28), and anger (12 items, range 0-48). Positive subscale includes vigor (8 items, range 0-32).
[11C]CURB decreases related to drug-related effects | 4 weeks
  Changes in drug-related assessment Addiction Research Center Inventory (ARCI) scores from baseline to post-nabilone (81 items, range 0-81) with higher score indicating greater drug-related effects.
[11C]CURB decreases related to drug-related effects | 1 week
  Changes in drug-related assessment Visual Analogue Scales (VAS) score from beginning of nabilone administration period to end of nabilone administration period. Score can range from a minimum of 0 (no pain) to a maximum of 10 (pain as bad as it could possibly be).
[11C]CURB related to blood measurements of endocannabinoids | 4 weeks
  Changes in blood measurements of endocannabinoids such as anandamide post-nabilone administration from baseline to post-nabilone.

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Boileau, PhD, Principal Investigator — Centre for Addiction and Mental Health; Stefan Kloiber, MD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
We will share and/or re-use the information that was already collected for this study with other researchers at CAMH or elsewhere, so it can be used in other studies to answer new or different scientific questions. We do not know what this research may be yet, but we think it will be related to future research on mental illness. The results of these studies will not be shared with participants from this study. Participants will not directly benefit from these future studies, but it is hoped that the research may help other people in the future. Any personal information that could identify participants will be removed or coded before the data is shared.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: June 2023 - indefinitely